CLINICAL TRIAL: NCT03875599
Title: Validation of the Pulmonary Rehabilitation Adapted Index of Self-Efficacy on Portuguese Respiratory Patients
Brief Title: Measuring Self-Efficacy on Portuguese Respiratory Patients on Pulmonary Rehabilitation
Acronym: PRAISEPort
Status: Completed | Type: Observational
Sponsor: University of Lisbon (Other)
Collaborators: Centro Hospitalar Lisboa Norte (Other); Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Principal Investigator, Catarina Santos, PhD student, Physiotherapist MSc, University of Lisbon
Other Study IDs: 46/17
Record Dates: First submitted 2019-03-11; First posted 2019-03-15 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Pulmonary Rehabilitation
Keywords: self-efficacy; instrument validity; PRAISE

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Pulmonary Rehabilitation — Respiratory Physiotherapy, Exercise Therapy, Patient Education

SUMMARY:
This study aimed to translate and adapt to portuguese an original british instrument useful to measure respiratory patients' self-efficacy specific to the context of Pulmonary Rehabilitation.

DETAILED DESCRIPTION:
Recent updates on Pulmonary Rehabilitation highlight the importance of patients' self-efficacy on long-term adherence to health-enhancing behaviors. The Pulmonary Rehabilitation Adapted Index of Self-Efficacy (PRAISE) is an adaptation of the General Self-Efficacy Scale. This study aimed to translate, culturally adapt and evaluate reliability and validity of PRAISE on Portuguese respiratory patients.Forward-backward translation and pilot testing were performed. Content validity was assessed by a multidisciplinary panel of expert judges. To evaluate reliability and validity, 150 respiratory outpatients on Pulmonary Rehabilitation participated on a cross-sectional study. Descriptive and reliability analyses, and exploratory factorial analysis using principal axis factoring, followed by oblique oblimin factor rotation were conducted to identify construct validity. IBM® SPSS® version 22 was used to perform statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute respiratory disease
* Patients with chronic respiratory disease
* Patients attending a hospital-based Pulmonary Rehabilitation program

Exclusion Criteria:

• Cognitive deficit for answering a questionnaire

Ages: 26 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 150 adults attending an outpatient Pulmonary Rehabilitation program based at Hospital Pulido Valente from Centro Hospitalar Universitário de Lisboa Norte, in Lisbon, Portugal.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2018-01-19 (Actual); Primary Completion 2018-11-23 (Actual); Study Completion 2018-11-23 (Actual)

PRIMARY OUTCOMES:
Patients' self-efficacy | 2 weeks
  Vincent and co-authors (2011) proposed the Pulmonary Rehabilitation Adapted Index of Self-Efficacy (PRAISE). The PRAISE tool is composed by a total of 15 items, combining 10 items from the General Self-Efficacy Scale (GSE) by Schwarzer and Jerusalem (1995), and 5 new specific items related to Pulmonary Rehabilitation. Each item is scored from 1 to 4 with a total range from 15 to 60, with higher scores indicating higher levels of self-efficacy. Araújo and Moura (2011) already validated a Portuguese version of the GSE, yet the assessment of self-efficacy remains to be explored on the Portuguese Pulmonary Rehabilitation setting. This study translated, culturally adapted and evaluated reliability and validity of PRAISE on Portuguese respiratory patients, with original author's permission. Hence, items 4, 7, 9, 12 and 15 were specific to Pulmonary Rehabilitation as proposed by PRAISE original authors, and the remaining items and answer key were in accordance with the portuguese GSE.

CONTACTS AND LOCATIONS:
Overall Officials: Catarina D Santos, MSc, Principal Investigator — University of Lisbon; Cristina Bárbara, PhD, Study Director — University of Lisbon
Locations (4):
- Portugal (4):
  - Instituto Nacional de Saúde Doutor Ricardo Jorge, Departamento de Epidemiologia, Lisbon
  - Universidade de Lisboa, Faculdade de Medicina, Instituto de Saúde Ambiental (ISAMB), Lisbon
  - Centro Hospitalar Universitário Lisboa Norte, Hospital Pulido Valente, Unidade de Reabilitação Respiratória, Lisbon
  - Instituto Politécnico de Lisboa, Escola Superior de Tecnologia da Saúde de Lisboa, Unidade de Ensino e Investigação em Psicologia e Sociologia, Lisbon

IPD SHARING:
Plan to Share IPD: No